CLINICAL TRIAL: NCT00958256
Title: Phase II Study of Bortezomib in Combination With Cyclophosphamide and Rituximab for Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Study of Bortezomib in Combination With Cyclophosphamide and Rituximab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0057; X05290; NCI-2009-01577 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-03

CONDITIONS: Mantle Cell Lymphoma; Lymphoma
Keywords: Mantle Cell Lymphoma; Lymphoma; Bortezomib; Velcade; Rituximab; Rituxan; Cyclophosphamide; Cytoxan; Neosar; Mesna; Mesnex; G-CSF; Filgrastim; Neupogen
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — Bortezomib; Rituximab; Cyclophosphamide; Mesna; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib with Cyclophosphamide and Rituximab (Experimental): Bortezomib 1.3 mg/m^2 intravenously (IV) on Days 1, 4, 8, and 11 of the cycle; Cyclophosphamide 300 mg/m^2 IV every 12 hours on Days 2, 3, and 4, and Rituximab 375 mg/m^2 IV on Day 1. Mesna 600 mg/m^2 for 3 days, G-CSF 5 micrograms/kg subcutaneously daily for 7 days after last dose of Bortezomib. Cycles repeated every 21 days for up to six cycles.
  Interventions: Drug: Bortezomib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Mesna; Drug: G-CSF

INTERVENTIONS:
Drug: Bortezomib — Bortezomib 1.3 mg/m^2 given intravenously over 3-5 seconds at the end of infusion of Rituximab on Day 1 of every cycle, then on Days 4, 8 and 11 of every cycle.
  Other Names: Velcade
Drug: Rituximab — 375 mg/m^2 given intravenously over 6-8 hours on Day 1 of every 21-day study cycle.
  Other Names: Rituxan
Drug: Cyclophosphamide — 300 mg/m^2 intravenously over 3 hours 2 times each day (6 hours total each day) on Days 2, 3, and 4 of every cycle
  Other Names: Cytoxan; Neosar
Drug: Mesna — 600 mg/m^2 intravenous continuous infusion (IVCI) over 24 hours daily for 3 days, 1 hour prior to Cyclophosphamide and complete by 12 hours after last dose of Cyclophosphamide.
  Other Names: Mesnex
Drug: G-CSF — 5 micrograms/kg subcutaneously daily starting 24-36 hours for 7 days after last dose of Bortezomib until granulocytes are more than 4 x 103/dl.
  Other Names: Filgrastim; Neupogen; Granulocyte-colony stimulating factor; GCSF

SUMMARY:
The goal of this clinical research study is to learn if bortezomib when given in combination with cyclophosphamide and rituximab can help to control mantle cell lymphoma. The safety of this drug combination will also continue to be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Bortezomib is designed to block a protein that plays a role in cell function and growth. This may cause cancer cells to die.

Cyclophosphamide is designed to interfere with the multiplication of cancer cells, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

Rituximab is designed to attach to lymphoma cells, which may cause them to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive all of the study drugs preferably through a central venous catheter (CVC) that will be left in place the entire time that you are receiving the study drugs. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. You will sign a separate consent form for this procedure, which will describe the procedure and the risk in more detail.

You will receive rituximab by vein over 6 hours on Day 1 of every 21-day study cycle.

You will receive bortezomib by vein over 3 to 5 seconds, after you have received rituximab on Day 1 of every cycle. You will also receive bortezomib on Days 4, 8, and 11 of every cycle.

You will receive cyclophosphamide by vein over 3 hours 2 times each day (6 hours total each day) on Days 2, 3, and 4 of every cycle. On these days, you will also receive mesna by vein non-stop. Mesna is a drug that protects the bladder from damage by chemotherapy drugs. It is used to decrease the risk of bleeding in the bladder.

You will receive G-CSF (filgrastim - a drug that is used to help build your white blood cell counts and prevent infections) as an injection under the skin starting 24-36 hours after you receive bortezomib. You will receive filgrastim 1 time each day until your white blood cell counts recover.

Study Visits:

At each study visit, you will be asked about how you are feeling and about any other drugs that you may be taking.

Throughout the study, blood (about 1 tablespoon each time) will be drawn 2-3 times a week for routine tests.

Within 2 days before each cycle, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will complete the questionnaire about nervous system side effects.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine tests.

After every 2 cycles, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will have a chest x-ray or CT scans to check the status of the disease. These scans may be of your head, neck, chest, stomach, and/or pelvis. The CT scan at Cycle 4 will only occur if the doctor thinks it is needed.
* Blood (about 5 teaspoons) will be drawn for routine tests.
* If your doctor thinks it is needed, you will have a bone marrow biopsy/aspirate to check the status of the disease.
* If your doctor thinks it is needed, you will have an ECHO or a multigated radionuclide angiography (MUGA) scan and/or an ECG.

You will have an exam of the colon (colonoscopy) to check the status of the disease after Cycle 2. Biopsy samples (about 3-6) of the colon will be taken during this exam to check the status of the disease.

After Cycles 2, 6, and/or 8, if your doctor thinks it is needed, you will have a positron emission tomography (PET) scan to check the status of the disease.

After Cycle 6, you will be taken off study if the disease is in "complete remission" (if the disease has disappeared). Otherwise, you may receive 2 more cycles of study treatment.

If you are receiving 2 more cycles, if colonoscopy was done after Cycle 2 and it showed lymphoma, you will have another colonoscopy after Cycle 6 and Cycle 8 to check the status of the disease. Biopsy samples (about 3-6) of the colon will be taken during this exam to check the status of the disease.

Length of Study:

You will receive the study drugs for up to 8 cycles (about 8 months). You will be taken off study early if the disease gets worse or intolerable side effects occur before Cycle 8, or if the disease is in complete remission after Cycle 6.

End-of-Treatment Visit:

After you have finished receiving the study drugs, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* You will complete the questionnaire about nervous system side effects.
* Your performance status will be recorded.
* You will have a chest x-ray or CT scans to check the status of the disease.
* Blood (about 5 teaspoons) will be drawn for routine tests.
* If your doctor thinks it is needed, you will have a bone marrow biopsy/aspirate to check the status of the disease.
* If your doctor thinks it is needed, you will have an ECHO or a MUGA scan and/or an ECG.

Follow-Up Visits:

After you have finished receiving the study drugs, you will have follow-up visits according to the following schedule:

* Every 3 months during Year 1 after treatment.
* Every 4 months during Year 2 after treatment
* Every 6 months during Years 3-4 after treatment.
* Every 12 months after Year 4 after treatment.

At each of the follow-up visits, the following tests and procedures will be performed:

* You will have a complete physical exam, including measurement of your weight and vital signs.
* You will complete the questionnaire about nervous system side effects.
* Your medical history will be recorded
* Your performance status will be recorded.
* Blood (around 1 tablespoon) will be drawn for routine tests.
* You will have a chest x-ray to check the status of the disease.
* You will have CT scans of the head, neck, chest, abdomen, and pelvis to check the status of the disease.
* If the doctor thinks it is needed, you will have a bone marrow aspirate/biopsy to check the status of the disease.

This is an investigational study. All of the drugs used in this study are FDA approved and commercially available for the treatment of various types of lymphoma. The use of this drug combination is investigational.

Up to 46 patients will take part in this multicenter study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis mantle cell lymphoma and its variants, excluding marginal zone and disease exclusively in the GI system. Patients should have measurable disease based on Cheson Criteria or Bone Marrow/tissue sample positive for mantle cell lymphoma. No prior therapy with a combination of bortezomib, cyclophosphamide and rituximab.
2. Patients with performance status of 2 or less (Zubrod).
3. Serum bilirubin <1.5 mg/dl and serum creatinine < 2.0 mg/dl unless due to lymphoma; absolute neutrophil count (ANC) >1000/mm^3 and platelets >100,000/mm^3 unless due to lymphoma.
4. Cardiac ejection fraction 50% or greater.
5. Ages 18 to 85.
6. Patients must be willing to receive transfusions of blood products.
7. Signed consent form.
8. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
9. Female subject is either post-menopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) from the time of signing the informed consent form through 30 days after the last dose of VELCADE, or agree to completely abstain from heterosexual intercourse.
10. Male subjects, even if surgically sterilized (ie, status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV) infection.
2. Central nervous system (CNS) involvement.
3. Patient has a platelet count of < 100 K (eg <30 x 10^9/L for studies with bortezomib alone) within 14 days before enrollment.
4. Patient has an absolute neutrophil count of ANC (eg <1.0 x 10^9/L for studies with bortezomib alone)> within 14 days before enrollment.
5. Patient has > 1.5 times Total Bilirubin
6. Patient has a calculated or measured creatinine clearance of < 20 mL/minute creatinine clearance (eg <20 mL/minute for studies with bortezomib alone) > within 14 days before enrollment.
7. Patient has >/= Grade 2 peripheral neuropathy within 14 days before enrollment.
8. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
9. Patient has hypersensitivity to bortezomib, boron or mannitol.
10. Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum Beta-human chorionic gonadotropin (Beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
11. Participation in clinical trials with other investigational agents not included in this trial, within 14 days the start of this trial and throughout the duration of this trial.
12. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
13. Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
14. Concurrent or previous malignancy whose prognosis is poor (< 90% probability of survival at 5 years).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Romaguera, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lee HJ, Romaguera JE, Feng L, Desai AP, Zhang L, Fanale M, Samaniego F, Hagemeister FB, Fayad LE, Rodriguez MA, Medeiros JL, Hartig K, Nomie K, Ahmed M, Badillo M, Ye H, Oki Y, Lin P, Nastoupil L, Westin J, Wang M. Phase II Study of Bortezomib in Combination with Cyclophosphamide and Rituximab for Relapsed or Refractory Mantle Cell Lymphoma. Oncologist. 2017 May;22(5):549-553. doi: 10.1634/theoncologist.2016-0328. Epub 2017 Apr 13. PMID 28408615
- See also: University of Texas MD Anderson Cancer Center Web Site — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 5, 2009 to March 28, 2013. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 22 participants enrolled, one participant was excluded from the trial before treatment.
Groups:
- Bortezomib With Cyclophosphamide and Rituximab: Bortezomib 1.3 mg/m^2 intravenously (IV) on Days 1, 4, 8, and 11 of the cycle; Cyclophosphamide 300 mg/m^2 IV every 12 hours on Days 2, 3, and 4, and Rituximab 375 mg/m^2 IV on Day 1. Mesna 600 mg/m^2 for 3 days, Granulocyte-colony stimulating factor (G-CSF) 5 micrograms/kg subcutaneously daily for 7 days after last dose of Bortezomib. Cycles repeated every 21 days for up to six cycles.
Period: Overall Study
Arm/Group | Bortezomib With Cyclophosphamide and Rituximab
Started | 21
Completed | 18
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: One participant of 21 participants was not treated and is therefore excluded from baseline demographics.
Arm/Group | Bortezomib With Cyclophosphamide and Rituximab
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 66 [48 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate to regimen defined as the percentage of number of complete response or partial response in total number of participants treated. The response assessed after the first 2 cycles. Response (complete and partial remission) according to International Workshop Response Criteria for Non-Hodgkin's Lymphoma: A complete response is the complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. A partial response is regression of measurable disease and no new sites of disease. Stable disease is failure to attain a complete response/partial response or progressive disease. A cycle is 21 days with 6-8 cycles administered depending on response.
Time Frame: Evaluation of disease after 2 cycles (approximately 6 weeks).
Population: Twenty-one patients were evaluable for response assessment (100%), of whom 16 responded (76%) thus reflected are the percentage of responses to total responders (i.e. 11 (52%) of total evaluable achieved a complete response).
Measure: Number; unit: percentage of participants
Arm/Group | Bortezomib With Cyclophosphamide and Rituximab
Number analyzed (Participants) | 21
percentage of participants
  Complete Response (CR) | 52
  Partial Response (PR) | 0
  Progressive Disease (PD) | 19
  Stable Disease (SD) | 5

ADVERSE EVENTS:
Time Frame: Adverse event collection performed with each cycle of chemotherapy every 21 days, up to 8 cycles with those who received at least one cycle considered assessable for adverse events. Overall study period: August 2009 to March 19, 2014.
Arm/Group | Bortezomib With Cyclophosphamide and Rituximab
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 21/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib With Cyclophosphamide and Rituximab (N=21)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 7 (13)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 12 (22)
Allergic rhinitis (Immune system disorders) | 6 (7)
Anorexia (Gastrointestinal disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3)
Arrhythmia supraventricular (Cardiac disorders) | 2 (2)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 11 (21)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilirubin increased (Blood and lymphatic system disorders) | 1 (1)
Blood glucose increased (Blood and lymphatic system disorders) | 18 (55)
Blood uric acid increased (Blood and lymphatic system disorders) | 11 (55)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bruising (General disorders) | 3 (3)
Cardiac General (Other) (Cardiac disorders) | 2 (2)
Chest wall pain (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Creatinine increased (Metabolism and nutrition disorders) | 5 (10)
Dehydration (Gastrointestinal disorders) | 2 (3)
Dermatology/Skin (Other) (Skin and subcutaneous tissue disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Dizziness (Nervous system disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 5 (6)
Fatigue (General disorders) | 16 (20)
Febrile neutropenia (Infections and infestations) | 1 (1)
Fever (Investigations) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal (Other) (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 19 (71)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3)
Hypertension (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Metabolism and nutrition disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 17 (125)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 12 (76)
Memory impairment (Nervous system disorders) | 1 (1)
Metabolic/Laboratory (Other) (Metabolism and nutrition disorders) | 20 (64)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal (Other) (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (18)
Neutrophil count decreased (Blood and lymphatic system disorders) | 19 (108)
Ocular/Visual (Other) (Eye disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 3 (4)
Pain (Other) (General disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 21 (148)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Pneumothorax (Infections and infestations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary (Other) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 10 (28)
Serum cacium decreased (Metabolism and nutrition disorders) | 9 (26)
Serum glucose decrease (Metabolism and nutrition disorders) | 3 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 7 (13)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium increased (Metabolism and nutrition disorders) | 3 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (11)
Serun potassium decreased (Metabolism and nutrition disorders) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes